CLINICAL TRIAL: NCT05877170
Title: Evaluation of the Analgesic and Anti-inflammatory Activities of a Nutraceutical Agent Containing PEA in the Management of Patients With Orofacial Pain, Both Neuropathic and Nociceptive in Nature
Brief Title: Impact of Palmitoylethanolamide (PEA) in the Management of Oro-facial Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal Researcher, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 121-25
Record Dates: First submitted 2023-05-15; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Oral-facial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEA (Experimental): PEA-containing nutraceutical agent in oral formulation
  Interventions: Dietary Supplement: Palmitoyletinolamide
- Placebo (Placebo Comparator): Patients treated with a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Palmitoyletinolamide — Taking a once-daily supplement containing PEA in an oral formulation (tablets), to be taken away from meals
  Arms: PEA
Drug: Placebo — Taking a placebo in an oral formulation (tablets), to be taken away from meals
  Arms: Placebo

SUMMARY:
Pain is the most common symptom faced by dentists, whether acute (pulpitis, acute periodontitis, post-surgical, etc.) or chronic (chronic periodontitis, muscle pain, TMJ disorders, BMS, OLP, etc.). The success of therapy depends on the reduction and management of pain. Therefore, over the past few years, the need has emerged, also in relation to the aging population, to analyze new molecules with pain-relieving activity and with low risk of inducing side effects and interactions with other drugs; capable of bringing about the reduction of oro-facial pain; and that lend themselves to prolonged use. Palmitoylethanolamide (PEA) is a bioactive lipid mediator similar to endocannabinoids (eCBs) that has been observed to have anti-inflammatory, analgesic, anticonvulsant, antimicrobial, antipyretic, antiepileptic, immunomodulatory, and neuroprotective activities.

The objective is to clinically study, through a clinical trial, the pain-relieving and anti-inflammatory properties of a PEA-containing nutraceutical agent in the management of patients with orofacial pain, both neuropathic and nociceptive in nature.

DETAILED DESCRIPTION:
A double-blind placebo-controlled study was conducted to evaluate the efficacy of Palmitoyletinolamide (PEA) and determine the statistical significance of its action.

40 patients with both acute and chronic orofacial pain were divided into two groups: study group given a nutraceutical agent containing PEA and a control group given a placebo. A three-month follow-up will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* good general health condition,
* presence of diffuse or localized oro-facial pain of nociceptive nature or postoperative pain,
* presence of diffuse or localized oro-facial pain of neuropathic nature for at least 1 month.

Exclusion Criteria:

* Allergies,
* debilitating systemic diseases,
* pregnancy status
* severe cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-08-12 (Estimated); Study Completion 2023-08-17 (Estimated)

PRIMARY OUTCOMES:
Reduction of oral-facial pain | 3 Months
  * The short-term and long-term effects of PEA on the management of neuropathic pain of the oro-facial district.
  * The short-term effects of PEA on the management of nociceptive pain of the oro-facial district.
  Visual Pain Analog Scale (VAS) will be used for pain assessment, in which the value 0 indicates no pain and the value 100 the maximum pain. The Oral Health Impact Profile Short For will be used to assess the impact of oral problems on quality of life, in which the presence or absence of physical pain, functional limitation, psychological distress, physical disability, physiological disability will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol